CLINICAL TRIAL: NCT07221110
Title: Effectiveness of Transcranial Magnetic Stimulation on Dysphagia in Patients With Parkinson's Disease: A Randomized Double-Blind Study
Brief Title: rTMS Treatment of Dysphagia in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Kübra Efe, Doctor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-70198063
Record Dates: First submitted 2025-10-22; First posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-09

CONDITIONS: Dysphagia; Parkinson's Disease (PD)
Keywords: rTMS; magnetic stimulation; Parkinson's disease; dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Transcranial Magnetic Stimulation; Exercise

STUDY DESIGN:
Intervention Model Description: Our patients will receive treatment at different frequencies on the same rTMS device.
Who Masked: Investigator
Masking Description: there is no
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 5 Hz (Experimental): Our patients in this arm will receive 10 sessions of treatment on the rTMS device. The device setting will be 5 Hz. All patients will also receive massako, shaker, triflo and cervical strengthening exercises. Our patients will be evaluated with FEES (Fiberoptic endoscopic swallowing evaluation) before, at the end of the treatment and at the 9th month controls in terms of the status of dysphagia.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Other: Exercise
- 10 Hz (Experimental): Our patients in this arm will receive 10 sessions of treatment on the rTMS device. The device setting will be 10 Hz. All patients will also receive massako, shaker, triflo and cervical strengthening exercises. Our patients will be evaluated with FEES (Fiberoptic endoscopic swallowing evaluation) before, at the end of the treatment and at the 9th month controls in terms of the status of dysphagia.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Other: Exercise

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — In our study, rTMS device was used to target the pharyngeal cortex for therapeutic purposes in patients with dysphagia diagnosed with Parkinson's disease. The most important point that distinguishes our study from other studies is that it aims to determine the effectiveness of rTMS treatment at high frequencies in the treatment of dysphagia. For this purpose, 5 Hz and 10 Hz treatments were applied to the patients from two different arms.
Other: Exercise — In our study, patients in both arms were given shaker, massako, cervical strengthening and triflo exercises.

SUMMARY:
The study was conducted with patients with dysphagia who were followed up with Parkinson's disease in the neurology and physical therapy rehabilitation departments. The study is a prospective, double-blind clinical intervention study. Patients were divided into two groups (5 Hz and 10 Hz) and received rTMS (repetitive transcranial magnetic stimulation) treatment. The pharyngeal cortex region was targeted in the intervention. Major aim in the treatment was to examine the difference in clinical response caused by the application of rTMS treatment at different frequencies.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease for more than two years
* Moderate-to-severe Parkinson's disease (Hoehn yahr 2-4)
* The patient describing dysphagia symptoms
* Patients being able to give informed consent.

Exclusion Criteria:

* İntracranial metallic device
* Cardiac pace-maker
* History of seizure
* İntracranial lesion on imaging
* Hydrocephalus
* Antipsychotic use
* Babinski positivity
* Berebellar symptoms
* Depression
* Dementia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
FEES evaluation | until two weeks after the start of treatment
  For the evaluation, a thin flexible nasopharyngoscope was passed through the nasal passage to visualize the pharynx and larynx. Food trials were performed for the swallowing assessment. For this purpose, patients were given water, nectar in volumes of 3-5-10-20 ml; 1 teaspoon (5 ml) of yogurt and 1 fish cracker. After the evaluation, early spillage, penetration, aspiration, and the presence/absence of residue in the pharyngeal wall/retrocricoid area/piriform sinus/vallekula were recorded. At the same time, the YALE-2016 vallekular residue scale, YALE-2016 piriform sinus residue scale, and penetration aspiration scale (PAS) scores were determined.
  YALE-2016 Vallekular/Piriform Sinus Residue Scale: This scale scores patients from 1 to 5 during flexible endoscopic examination based on the amount of residue in the vallekula and piriform sinus: none/trace/mild/moderate/severe.
  PAS: This scale rates patients from 1to5 based on aspiration/penetration and the presence of a protective reflex
Swallowing Assessment Form: | up to two weeks after the start of treatment
  The form records data on patients' age, gender, duration of Parkinson's disease, duration of dysphagia, history of pneumonia, Hoehn-Yahr stage, type of nutrition, dysphagia with solid food, dysphagia with semi-solid food, dysphagia with liquid food, sensation of food getting stuck in the throat, sensation of choking, and need to clear the throat.
Functional Oral Intake Scale (FOIS): | until two weeks after the start of treatment
  Oral intake in patients; no oral intake (1), minimal attempt at solid-liquid food, dependent on tube feeding (2), continuous solid and liquid oral intake, but dependent on tube feeding (3), total oral diet of uniform consistency (4), total oral diet of varying consistencies, but requiring special preparation or compensation (5), total oral diet of varying consistencies, not requiring special preparation, but with specific food limitations (6), total oral diet without restrictions (7).
Functional Swallowing Scale (FSS): | until two weeks after the start of treatment
  This scale assesses patients' daily dysphagia symptoms and associated weight loss. Patients are classified as normal function and asymptomatic (0), normal function with episodic or daily dysphagia symptoms (1), abnormal function compensated by significant dietary modifications (2), and abnormal function with decompensation, with <10% weight loss in the last 6 months due to dysphagia or coughing/ choking/aspiration during daily meals (3), severe decompensated abnormal function with >10% weight loss in the last 6 months due to dysphagia/severe aspiration/non-oral feeding for most foods (4), non-oral feeding for all foods (5).
Swallowing Function Screening Test (EAT-10): | until two weeks after the start of treatment
  An EAT-10 score of 3 or higher indicates abnormality. This test can be used to determine the initial severity of dysphagia in individuals with various swallowing disorders or to monitor treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Eyigor, Study Director — Ege University Hospital
Locations (1):
- Ege University Hospital, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
For the purpose of protecting personal data, individual participant data will not be shared.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT07221110/Prot_SAP_000.pdf
  • Informed Consent Form (2025-10-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT07221110/ICF_001.pdf